CLINICAL TRIAL: NCT05911282
Title: N-acetylcysteine Reduces Acetaldehyde Levels in Binge Alcohol Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miran Brvar, Head of Centre for Clinical Toxicology and Pharmacology, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20200175
Record Dates: First submitted 2023-05-29; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ethanol Intoxication
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC (Experimental): NAC group was given 1.2 g of N-acetylcysteine before and 1.2 g after drinking alcohol
  Interventions: Drug: N Acetylcysteine
- PLACEBO (Placebo Comparator): Placebo group was given lemon juice before and after drinking alcohol
  Interventions: Other: Lemon juice

INTERVENTIONS:
Drug: N Acetylcysteine — The study began at 7 pm, when the volunteers in NAC group drank the contents of a numbered cup with NAC (1.2 g of NAC). At 9 pm, they were given the second cup with 1.2 g of NAC corresponding to their randomized number.
  The cups with pure substance NAC were prepared and numbered by the physician not attending the drinking just before the study.
  Other Names: NAC
  Arms: NAC
Other: Lemon juice — The study began at 7 pm, when the volunteers in placebo group drank the contents of a numbered cup with lemon juice. At 9 pm, they were given the second cup with lemon juice corresponding to their randomized number.
  The cups with lemon juice were prepared and numbered by the physician not attending the drinking just before the study.
  Other Names: placebo
  Arms: PLACEBO

SUMMARY:
Alcohol hangover (veisalgia) is a fairly common phenomenon. The pathogenesis of veisalgia is not understood and treatment has not yet been established. Occasionally, students take N-acetylcysteine (NAC) before binge drinking to alleviate hangover. The aim of the study was to evaluate the effect of NAC on serum levels of electrolytes, enzymes, acetaldehyde, oxidative stress biomarkers and symptoms of veisalgia in binge drinking. In this randomised double-blind placebo-controlled study, healthy students were randomly assigned into two groups, one receiving NAC and the other placebo. Blood samples were taken before drinking, 30 minutes after 1.5-hour-long drinking and in the subsequent morning. Serum levels of electrolytes, urea, enzymes, ethanol, acetaldehyde, 8-Hydroxydeoxyguanosine (8-OHdG) and N-epsilon-hexanoyl-lysine were measured. The participants completed the Acute Hangover Severity Scale (AHSS) based on symptoms.

DETAILED DESCRIPTION:
On the study day, the participants met at the study location with the investigator at 6.pm. In the beginning they all ate two pizza slices. They filled out a pre-drinking evaluation form about veisalgia (score 1 - 10) and specific symptoms (score 1 - 10). They performed a breath alcohol test with Dräger Alcotest 6820 to exclude volunteers who had been drinking before the study. The registered nurses took blood samples before drinking.

Volunteers were randomly assigned into two groups, one receiving NAC (1.2 g before and 1.2 g after drinking alcohol), and the other placebo. Each participant received an identification number, randomisation was done by a computer. The study began at 7 pm, when they drank the contents of a numbered cup with NAC or placebo corresponding to their number. The researchers and volunteers on the scene were not aware which cups contain NAC or placebo. Afterwards they drank 40 %, v/v, gin mixed with tonic according to the participant's preferences. The drinking was calm. They were mostly sitting and did not participate in any physical activity such as dancing. No other legal or illegal substances or medications were taken during the study.

The drinking ended at 8.30 pm. The nurses took the second blood sample 30 minutes after 1.5-hour-long drinking. The volunteers also performed the second breath alcohol test.

At 9 pm, they were given the second cup with 1.2 g of NAC or placebo corresponding to their randomized number. The latest one hour after the second blood sample was taken all the participants went to sleep.

In the next morning at 6 am (9 hours after drinking) the third blood sample was taken in all volunteers. They performed the third breath alcohol test and filled out a post-drinking form about veisalgia (score 1 - 10), specific symptoms (score 1 - 10), and Alcohol Hangover Severity Scale (AHSS).

ELIGIBILITY:
Inclusion Criteria:

* medical students, who regularly attend social gatherings where alcohol is consumed and had already experienced the symptoms of hangover.
* healthy
* not pregnant
* without any chronic diseases
* not taking any medications.
* signed informed consent.

Exclusion Criteria:

* drinking after the end of the study
* taking any other psychoactive substances or took other measures that supposedly could alleviate the hangover symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Alcohol Hangover Severity Scale | next morning after drinking (at 6 am; 9 hours after drinking)
  In the next morning after drinking (at 6 am; 9 hours after drinking) the volunteers filled out a standardised questionnaire Alcohol Hangover Severity Scale (AHSS), which includes twelve symptoms correlating with veisalgia: palpitation, sweating, confusion, apathy, abdominal pain, shivering, dizziness, nausea, clumsiness, concentration problems, thirst and fatigue.
  Every symptom was graded on the scale from 0 to 10 points, where 0 point meant the absence of the symptom and 10 points the extreme severity of the symptom.
  The result of the AHSS questionnaire was calculated for every participant as the average number of points from all of the 12 symptoms (minimum average value was 0 points and maximum 10 points).
Change in acetaldehyde level after drinking compared to the baseline value | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of acetaldehyde in blood samples
Change in serum oxidative biomarker level after drinking compared to the baseline value | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of 8-Hydroxydeoxyguanosine and N-epsilon-hexanoyl-lysin in blood samples

SECONDARY OUTCOMES:
Change in serum ethanol level after drinking compared to the baseline value | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of ethanol in blood samples
Change in serum sodium levels after drinking compared to the baseline | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of serum sodium in blood samples
Change in serum potassium levels after drinking compared to the baseline | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of serum potassium in blood samples
Change in serum urea levels after drinking compared to the baseline | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of serum urea in blood samples
Change in serum creatinine levels after drinking compared to the baseline | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of serum creatinine in blood samples
Change in serum creatinine kinase levels after drinking compared to the baseline | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of serum creatinine kinase in blood samples
Change in serum lactate dehydrogenase levels after drinking compared to the baseline | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of serum lactate dehydrogenase in blood samples
Change in serum aspartate and alanine aminotransferase levels after drinking compared to the baseline | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of serum aspartate and alanine aminotransferase in blood samples
Change in serum gamma glutamyl transferase levels after drinking compared to the baseline | before drinking (at 7 pm), within 30 minutes after 1.5 hour long drinking (at 9 pm) and in the next morning after drinking (at 6 am, 9 hours after drinking)
  Quantification of serum gamma glutamyl transferase in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Miran Brvar, MD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No